CLINICAL TRIAL: NCT00395707
Title: Phase I Study Of Intravitreal Ranibizumab (Lucentis) For The Treatment Of Stage 1 And 2 Retinal Angiomatous Proliferations
Brief Title: Study To Determine Safety/Efficacy of Lucentis For Treatment Of Retinal Angiomatous Proliferation Secondary To Age Related Macular Degeneration
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: The National Retina Institute (Other)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: T. Mark Johnson, MD, National Retina Institute
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: FVF3423s
Record Dates: First submitted 2006-11-01; First posted 2006-11-03 (Estimated); Last update posted 2009-02-09 (Estimated); Status verified 2009-02

CONDITIONS: Macular Degeneration
Keywords: Macular Degeneration; Age Related Macular Degeneration; Retinal Angiomatous Proliferations
MeSH Terms: conditions — Macular Degeneration | interventions — Ranibizumab

STUDY DESIGN:
Who Masked: Participant

ARMS (2):
- 1 (Active Comparator): Lucentis 0.3mg/0.05 ml
  Interventions: Drug: Lucentis; Drug: Ranibizumab; Drug: Ranibizumab (Lucentis)
- 2 (Active Comparator): Lucentis 0.5mg/0.05 ml
  Interventions: Drug: Lucentis; Drug: Ranibizumab; Drug: Ranibizumab (Lucentis)

INTERVENTIONS:
Drug: Lucentis — 0.3mg/0.05 ml or 0.5mg/0.05 ml
  Other Names: Ranibizumab
Drug: Ranibizumab — 0.3mg/0.05 ml or 0.5mg/0.05 ml
  Other Names: Lucentis
Drug: Ranibizumab (Lucentis) — 0.3mg/0.05 ml intravitreally
  Other Names: Ranibizumab; Lucentis
  Arms: 1
Drug: Ranibizumab (Lucentis) — 0.5mg/0.05 ml
  Other Names: Ranibizumab; Lucentis
  Arms: 2

SUMMARY:
The primary objective of this study is to determine the safety & efficacy of ranibizumab for the treatment of retinal angiomatous proliferation secondary to age related macular degeneration.

DETAILED DESCRIPTION:
This study will be a phase I/II open label interventional case series. Twenty patients with retinal angiomatous proliferation will be randomized to receive intravitreal ranibizumab at a dose of 0.3mg/0.05 ml or 0.5mg/0.05 ml. Patients will receive ranibizumab via a pars plana injection on a monthly basis for a total duration of therapy of 12 months. Patients will be followed for a complete 12-month treatment course.

ELIGIBILITY:
Inclusion Criteria:

* Ability to provide written informed consent and comply with study assessments for the full duration of the study.
* Age > 50 years
* Definite characteristic signs of age related macular degeneration including drusen
* Presence of retinal angiomatous proliferation as determined by clinical signs (intra retinal hemorrhage, retinal edema, cystic retinal edema) and angiography (occult leakage on fluorescein angiography, hot spot on static ICG, visible RAP lesion of high speed ICG)

Exclusion Criteria:

* Prior treatment with verteporfin, external-beam radiation therapy, or transpupillary thermotherapy in the study eye (predominantly classic CNV can however only be included if the subject had up to 3 prior PDT treatments)
* Treatment with verteporfin in the non-study eye less than 7 days preceding Day 0
* Previous participation in a clinical trial (for either eye) involving anti angiogenic drugs (pegaptanib, ranibizumab, anecortave acetate, protein kinase C inhibitors, etc.)
* Previous subfoveal focal laser photocoagulation involving the foveal center in the study eye
* Laser photocoagulation (juxtafoveal or extrafoveal) in the study eye within 1 month preceding Day 0
* History of vitrectomy, submacular surgery, or other surgical intervention for AMD in the study eye
* Previous participation in any studies of investigational drugs within 1 month preceding Day 0 (excluding vitamins and minerals)

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2005-08; Primary Completion 2008-04 (Actual); Study Completion 2008-04 (Actual)

PRIMARY OUTCOMES:
Proportion of patients with stabilization of visual acuity, vision loss of < 15 letters | 2 years
Proportion of subjects who gain at least 15 letters in the best corrected visual acuity score at 6 and 12 months compared to baseline | 12 months
Incidence and severity of ocular adverse events | 12 months
Incidence and severity of non-ocular adverse events | 12 months
Changes in vital signs | 12 months

SECONDARY OUTCOMES:
Assess the systemic and local safety of ranibizumab (0.3mg or 0.5mg) in patients with RAP lesions | 12 months
Assess the impact of ranibizumab (0.3mg or 0.5mg) on time to improvement in retinal thickness by OCT | 2 years
Assess the impact of ranibizumab (0.3mg or 0.5 mg) on leakage from RAP lesions by Fluorescein angiography | 2 years
Static / high speed ICG appearance to assess the impact of ranibizumab (0.3mg or 0.5mg) on persistence / recurrence of RAP lesion and monitor for development of retinal-choroidal anastomoses | 2 years
Assess the impact of ranibizumab (0.3mg or 0.5mg) on development of retinal-choroidal anastomoses as determined on clinical examination and high speed ICG | 2 years
Assess the impact of ranibizumab (0.3mg or 0.5mg) on development of subretinal fibrosis as determined by clinical examination | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Thomas M Johnson, MD, Principal Investigator — National Retina Institute
Locations (2):
- United States (2):
  - National Retina Institute, Chevy Chase, Maryland
  - National Retina Institute, Towson, Maryland